CLINICAL TRIAL: NCT04682600
Title: The Sonic Incytes Liver Incytes System, Evaluation of Liver Fibrosis and Steatosis Versus MRE and MRI PDFF
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Sonic Incytes (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: SI-CLIN-02
Record Dates: First submitted 2020-10-20; First posted 2020-12-24 (Actual); Last update posted 2022-12-09 (Actual); Status verified 2022-12

CONDITIONS: Non-Alcoholic Fatty Liver Disease (NAFLD); Non-Alcoholic Steatohepatitis (NASH); Liver Fibroses; Liver Steatoses
Keywords: NASH; NAFL; NAKLD; Liver; Elastography; Ultrasound
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease; Liver Cirrhosis; Fatty Liver

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Open-label (Experimental): Volunteers who have agreed to participate in the study will have their liver scanned using the FibroScan, VE (Liver Incytes System) and MRE techniques.
  Interventions: Device: Liver Incytes System

INTERVENTIONS:
Device: Liver Incytes System — The Liver Incytes System uses the Shear Wave Absolute Vibro-Elastrography (S-WAVE) method. The imaging procedure of the Liver Incytes system is similar to a traditional ultrasound scanning procedure or FibroScan, in which the patient is asked to lie supine on an examination bed, with the operator seated next to them. A vibration source is placed under the patient, between the patient and the bed to induce shear waves in the liver. Ultrasound imaging through the patient ribs is used to track the displacements of these waves. Through tracking of the displacements, the shear wave velocity and tissue stiffness can be calculated. The use of volumetric multi-frequency imaging increases the amount of liver scanned
  Other Names: MRE; MRI PDFF; Fibroscan

SUMMARY:
The main purpose of this study is to compare the effectiveness of various non-invasive elastography techniques at determining liver stiffness measures in human subjects. Specifically, the investigators are comparing MRE and FibroScan to Vibroelastography (VE, Liver Incytes System). These techniques are used to measure stiffness in the liver.

DETAILED DESCRIPTION:
The Liver Incytes system allows for full visualization of the liver with the low cost and portability of ultrasound. It is an adjustable multi-frequency technique, which can show large areas of the organ as volumetric elasticity maps. The device uses the Shear Wave Absolute Vibro-Elastography (S-WAVE) method.

The primary objective of the study is to determine the relationship between the elasticity results from Liver Incytes and those of MR Elastography. In addition to stiffness measurements, the relationship between the Liver Incytes attenuation measurements and MR-PDFF will also be evaluated.

As secondary objectives, the ability of Liver Incytes to correctly stage patients using MRE as the standard (unless biopsy is available), looking specifically at the ability to measure mild and advanced fibrosis.

In additional to performance objectives, the safety, tolerability and usability of the device will be assessed.

This is a prospective, open label, validation study of the Liver Incytes system in comparison to MR results (as gold standard) in patients with liver disease or suspected liver disease. Approximately 100 subjects may be enrolled in this study which will take place at clinical centers across Canada and the United States. Study participants should be distributed primarily across the 4 stages of fibrosis, with secondary consideration of the three stages of steatosis.

The study is comprised of: Screening Period (up to 28 days) and Data Collection Period. There are no safety follow-up visits in this study.

* Screening Period (-28 days to Prior to Imaging (Fibroscan, Liver Incytes, MRE)): during the screening phase, participants will provide written informed consent before undergoing procedures to determine study eligibility.
* Data Collection Period (variable duration): Study participants will attend a study visit on Day 1 and may attend an optional visit within 28 days of the initial/Day 1 visit.

The total duration of study participation will vary from approximately 2 weeks to approximately 8 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Adults, 19-75 years old
* Healthy volunteers or Patients with evidence of NAFLD such as one of the following:

Previous liver biopsy consistent with NAFLD OR

Evidence of hepatic steatosis on non-invasive assessment by one or more of the following criteria:

* Abdominal ultrasound within 12 months
* MRI-PDFF (greater than 12%) within 12 month
* FibroScan CAP score > 230 dB/m within 12 months OR At least 2 criteria for metabolic syndrome and increased stiffness on FibroScan (>8kPa) within 12 months
* Able to understand the informed consent form, study procedures and willing to participate in study
* If female and of child bearing potential, must agree to practice a highly effective contraception method.

Exclusion Criteria:

* Active viral hepatitis

  a. Patients with cured HCV (those with history of treatment and have Sustained Viral Response for 12 weeks (SVR12)) or controlled HBV with no viral detected for more than 6 months are eligible
* Decompensated cirrhosis (history of ascites, encephalopathy, or variceal bleeding)
* ALT or AST > 5 x ULN on historical blood work within the past 3 months
* BMI greater than 40 kg/m2 (or using cutoff based on MRI)
* Other known causes of chronic liver disease
* Individuals with history of persistent ethanol abuse (alcohol consumption > 20g etoh/day for women, > 40 g etoh/day for men)
* Individuals with surgically removed gallbladder
* Pregnant or planning to become pregnant while enrolled in this study
* Other conditions which would exclude patients from entering an MRI

Ages: 19 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 164 (Actual)
Dates: Start 2020-10-21 (Actual); Primary Completion 2022-11-01 (Actual); Study Completion 2023-07-01 (Estimated)

PRIMARY OUTCOMES:
Elasticity measurements comparison between Liver Incytes MR Elastography | 12 months
  Elasticity measurements (kPa) from the Liver Incytes system and the MR system will be compared to determined whether the reported stiffness of the tissue (mean and 95% confidence intervals) are equivalent by concordance correlation coefficient and 95% confidence intervals.
Determination of Liver Incytes' discriminatory ability of liver stiffness as measured by fibrosis staging | 12 months
  Liver Incytes liver stiffness values will be compared to values obtained using MRE to determine the cutoff values for the Liver Incytes System for each level of fibrosis staging. For each stage of fibrosis as defined by MRE, Area Under the Receiver Operating Curve (AUROC) for Liver Incytes elasticity will be calculated and the cutoff maximizing the sensitivity and specificity will be determined.

SECONDARY OUTCOMES:
Attenuation measurements comparison between the Liver incytes System and MRI Proton Density Fat Fraction | 12 months
  Attenuation measurements (dB/m) from the Liver Incytes System and MRI proton density fat fraction will be compared to determine whether they are equivalent by concordance correlation coefficient and 95% confidence intervals
Comparison between Liver Incytes' and FibroScan's fibrosis staging capabilities | 12 months
  Compare the discriminatory ability of Liver Incytes' and FibroScan's elasticity (kPa) measurements in determining different stages of fibrosis using MRE as gold standard.
  For each stage of fibrosis, a Receiver Operating Curve will be constructed using the corresponding FibroScan measurements, and the Area Under the Receiver Operating Curve (AUROC) will be compared to the result from Liver Incytes.
Comparison between Liver Incytes' and FibroScan's steatosis staging capabilities | 12 months
  Compare the discriminatory ability of Liver Incytes' and FibroScan's attenuation measurements (dB/m) in determining different stages of steatosis using MRE as gold standard.
  For each stage of steatosis, a Receiver Operating Curve will be constructed using the corresponding FibroScan measurements, and the Area Under the Receiver Operating Curve (AUROC) will be compared to the result from Liver Incytes.
Incidence of and Device Deficiencies | 12 months
  The frequency of device deficiencies and failures will be described based on events reported
Incidence of Adverse Events | 12 Months
  Descriptive statistics including frequency and severity of all reported adverse events.

OTHER OUTCOMES:
Identification of cases in which FibroScan may overestimate or underestimate liver stiffness | 12 months
  The elasticity (kPa) output from Liver Incytes, FibroScan, and MRE/PDFF will be used to identify and compare the cases in which the measurements do not match. Descriptive statistics regarding the populations in which the FibroScan systematically over or underestimates compared to MRE/MRI PDFF and the corresponding results from Liver Incytes
Identification of cases in which FibroScan may overestimate or underestimate fat content | 12 months
  The attenuation (dB/m) output from Liver Incytes, FibroScan, and MRE/PDFF will be used to identify and compare the cases in which the measurements do not match. Descriptive statistics regarding the populations in which the FibroScan systematically over or underestimates compared to MRE/MRI PDFF and the corresponding results from Liver Incytes
Liver Incytes System User Experience Survey | 12 months
  Descriptive statistics such as N, proportion, mean, median, SD, and range will be calculated for the composite score of the User Experience Survey, based on the modified System Usability Scale (mSUS). Descriptive statistics such as N, proportion, mean, median, SD, and range will be calculated for each question in the User Experience Survey and Liver Incytes Session Questionnaire.
  The modified SUS yields a single number representing a composite measure of the overall usability of the system being studied. It is composed of 10 questions, 5 positive in nature, and 5 negative. The score ranges from 0 to 6 and higher scores may mean a better or worse outcome depending on whether the question is positive or negative.
Liver Incytes System Inter-user Elasticity Variability | 12 months
  For subjects who participate in the optional additional visit, inter-user device variability, if applicable, will be assessed by comparing reported elasticity (kPa). Variance for each measurement will be calculated.
Liver Incytes System Inter-user Attenuation Variability | 12 months
  For subjects who participate in the optional additional visit, inter-user device variability, if applicable, will be assessed by comparing reported attenuation (dB/m). Variance for each measurement will be calculated.
Liver Incytes System Intra-Subject Variability | 12 months
  For subjects who participate in the optional additional visit, intra-subject variability will be assessed by comparing reported elasticity (kPa). Variance for each measurement will be calculated.

CONTACTS AND LOCATIONS:
Locations (1):
- Beth Israel Deaconess Medical Centre, Boston, Massachusetts, United States